CLINICAL TRIAL: NCT06719037
Title: Efficacy and Safety of Endo-Surgi Plus Endoscopy, UBE Endoscopy, and Microdiscectomy Decompression Techniques for the Treatment of Lumbar Spinal Stenosis: A Prospective Multicenter Study
Brief Title: Comparision of Endoscopic Discectomy and Microdiscectomy for the Treatment of Lumbar Spinal Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KYLL-202208-046-1
Record Dates: First submitted 2024-11-18; First posted 2024-12-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Microdiscectomy; Endoscopic; Unilateral Biportal Endoscopic; Endo-surgi Plus endoscopy; ODI; Complication; CK-MB
MeSH Terms: conditions — Spinal Stenosis | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endo-Surgi Plus endoscopic group (Experimental)
  Interventions: Procedure: Endo-Surgi Plus endoscopic surgery
- Unilateral biportal endoscopic group (Experimental)
  Interventions: Procedure: Unilateral biportal endoscopic surgery
- Microdiscectomy group (Active Comparator)
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: Endo-Surgi Plus endoscopic surgery — Endo-Surgi Plus endoscopic surgery, as a new type of percutaneous endoscopic lumbar discectomy (PELD), features a larger working channel and represents an optimized single-channel endoscopic technique. However, it still has the limitations inherent in single-channel endoscopy.
  Arms: Endo-Surgi Plus endoscopic group
Procedure: Unilateral biportal endoscopic surgery — Unilateral biportal endoscopic discectomy (UBE) is characterized by its separate endoscopic and working channels, and the ability to use traditional open instruments, making it a convenient and versatile technique. It is a commonly used spinal endoscopic surgery in clinical practice.
  Arms: Unilateral biportal endoscopic group
Procedure: Microdiscectomy — Microdiscectomy (MD) is a mature minimally invasive technique that uses a microscope to treat lumbar spinal stenosis. As early as 1999, prospective randomized controlled studies confirmed that it has equally excellent clinical efficacy compared to open surgery, with less surgical trauma. It is currently the classic minimally invasive surgical approach for treating lumbar spinal stenosis.
  Arms: Microdiscectomy group

SUMMARY:
The purpose of this study is to conduct a multicenter comparison of the clinical efficacy of Endo-Surgi Plus endoscopic technique, UBE endoscopic technique, and microdiscectomy technique in the treatment of lumbar spinal stenosis, and to compare the differences in the incidence of complications, surgical trauma, and other aspects among the three surgical techniques for the treatment of lumbar spinal stenosis.

Each group of patients received either Endo-Surgi Plus endoscopy, UBE, or microdiscectomy decompression through the Quadrant channel. All patients were routinely administered low-dose hormones, dehydrating agents, and neurotrophic drugs postoperatively. Patients were required to strictly avoid strenuous activities and heavy lifting in the lumbar region for three months after surgery. Upon discharge, patients were provided with the same lumbar and back muscle rehabilitation exercises and other postoperative recovery-related discharge education. Each group of patients was followed up for at least one year, with follow-up including outpatient visits, physical examinations, questionnaire scoring, and necessary auxiliary examinations.

Both two endoscopic surgeries, as surgical techniques that have been used in clinical practice for many years, have their efficacy confirmed by various studies. The investigator proposes that these two techniques may have similar clinical efficacy to microdiscectomy, while also offering the advantage of being less invasive. The aim of this study is to validate these assumptions. At the same time, there may be some differences between the two endoscopic surgeries that require further verification.

DETAILED DESCRIPTION:
The lumbar spine is the part of the spine that bears the most weight, consisting of five vertebrae. Each vertebra is connected by an intervertebral disc, and together they form a barrier to protect the spinal cord nerves within the spinal canal. Lumbar spinal stenosis refers to the reduction of space within the lumbar spinal canal, which compresses the spinal cord or nerve roots, leading to a series of symptoms. Depending on the cause, lumbar spinal stenosis is mainly divided into congenital lumbar spinal stenosis, which is due to abnormal development of the spinal canal, and acquired lumbar spinal stenosis, which is caused by degenerative changes such as lumbar disc degeneration and joint process hyperplasia. Lumbar spinal stenosis is a common cause of low back and leg pain, with a reported incidence rate as high as 11% in the general population and 19.4% in those over 60 years old, with a trend of increasing with age. With the aging of the population, the incidence of lumbar spinal stenosis is also on the rise.

The treatment of lumbar spinal stenosis mainly includes conservative treatment and surgical treatment. For patients whose symptoms severely affect their lives and do not respond well to conservative treatment, surgery should be performed as soon as possible to relieve nerve compression. The main goal of surgical treatment for lumbar spinal stenosis is to relieve nerve compression, stabilize the spine, and restore the normal volume of the spinal canal. Although traditional posterior lumbar decompression surgery can achieve definite decompression effects, it has issues such as severe destruction of posterior column structures and large surgical trauma. Minimally invasive techniques are a hot topic in various clinical fields, and microdiscectomy (MD) through a minimally invasive channel is a mature minimally invasive technique for treating lumbar spinal stenosis. As early as 1999, prospective randomized controlled studies confirmed that it has the same excellent clinical efficacy as open surgery but with less surgical trauma. It has now become a classic surgical method for treating lumbar spinal stenosis, with related articles published in the top spinal clinical journal JBJS.

In recent years, with the development of new equipment, endoscopic techniques have been gradually applied to the treatment of lumbar spinal stenosis. Unilateral biportal endoscopic discectomy (UBE) has the characteristics of convenient operation and flexibility because its endoscopic channel and working channel are separate and can use traditional open instruments. It can achieve good decompression effects and has been widely used in various medical centers. Percutaneous endoscopic lumbar discectomy (PELD), as a new generation of endoscopic technique, has less surgical trauma and shorter operation time. It has also been successfully applied to the clinical treatment of lumbar spinal stenosis and achieved good results. However, due to the limitations of the single-endoscopic channel field of view, its learning curve is steep, the surgical difficulty is high, and it is difficult to achieve complete decompression for bilateral spinal stenosis or dorsal nerve root compression. The efficiency of dealing with bony stenosis structures during surgery is low, leading to longer operation time and increased risk of nerve root and dural sac injury. Many clinical studies have compared the advantages and disadvantages of endoscopic techniques with traditional minimally invasive techniques and different endoscopic techniques, concluding that various endoscopic techniques can achieve surgical efficacy similar to traditional techniques with the advantages of less surgical trauma and faster postoperative recovery. Guilherme et al. believe that PELD has similar clinical efficacy to MD, but MD is superior for complex foraminal stenosis. In addition, a review by Ohyuk et al. suggests that UBE has better clinical efficacy and a lower complication rate compared to MD or PELD. However, most of these studies are small-scale, single-center, and retrospective, and the conclusions lack high-quality evidence support.

In recent years, single-channel decompression techniques under endoscopy have developed rapidly, especially large-channel endoscopes and related tools, which have significantly improved work efficiency and surgical safety. Many hospitals and medical research centers have introduced the Endo-Surgi Plus working channel, which has a larger working tube than traditional endoscopes, making it easier to treat certain types of lumbar disc herniation and lumbar spinal stenosis, further optimizing spinal endoscopic surgery techniques for lumbar spinal stenosis.

With the development of surgical instruments and approaches, these three minimally invasive spinal canal decompression techniques can effectively relieve pain symptoms in patients with various types of lumbar spinal stenosis. Compared with traditional open surgery, these techniques have reduced operation time, intraoperative blood loss, and postoperative pain. However, there are slight differences in the degree of trauma and ease of operation among these three techniques. Currently, there is still a lack of prospective validation of the clinical efficacy of these surgical techniques internationally, and the advantages and disadvantages of different endoscopic surgeries compared to traditional fenestration surgery.The purpose of this study is to conduct a multicenter comparison of the clinical efficacy of Endo-Surgi Plus endoscopic technique, UBE endoscopic technique, and microdiscectomy technique in the treatment of lumbar spinal stenosis.

Subjects were randomly divided into the Endo-Surgi Plus endoscopy group, the UBE group, and the fenestration group through the Quadrant channel. Randomization (1:1:1 grouping) was conducted within 2 weeks before surgery. Investigators used a block randomization design, stratified by 23 hospitals, with non-competitive enrollment between hospitals. The blocks were kept as small as possible (randomly selected block sizes of 3 and 6) to ensure that each hospital performed a similar number of all three types of surgeries. The computer-generated allocation output was sent via email to the local study coordinators (CRC), who did not participate in patient recruitment or treatment.

Due to the nature of the interventions, double blinding was not feasible. Randomization of patients aimed to reduce potential biases in preoperative planning and patient treatment. Throughout the study, outcome assessors and data analysts remained blinded to reduce biases in clinical outcome assessment and data analysis. Patients were informed that no treatment regimen was recorded as superior to another.

Determination of Sample Size: This study is a randomized controlled trial, with the postoperative 1-year ODI score of the subjects as the main outcome indicator. The trial required 324 patients to be included in total, with 80% statistical power to detect a difference of at least 12 points in ODI scores between treatment groups at a significance level of 0.05.Investigators conservatively chose a difference of 12 points because the U.S. Food and Drug Administration suggests that a 15-point reduction in ODI score indicates a minimally important improvement after spinal fusion surgery. Investigators conservatively set the standard deviation of the ODI score to 18, and estimated a dropout rate of 15%. Finally investigators used PASS to estimate that the trial would need to include a total of 324 patients.

Statistical and Analytical Plan: Patients who underwent the designated surgery and completed at least one year of follow-up were included. For continuous data that met normal distribution, analysis of variance (ANOVA) and post-hoc tests were used to compare differences among the three treatment groups; otherwise, the Kruskal-Wallis H-test was applied. Categorical variables were analyzed using chi-square or Fisher's exact test (expressed in numbers and percentages) to compare baseline characteristics among groups.

A mixed-effects model for repeated measures was used to compare changes in ODI and SF-36 scores relative to baseline across groups. Considering the correlation of repeated measures within patients, an unstructured covariance matrix was specified. The model included fixed effects for treatment (Endo-Surgi Plus endoscopy, UBE, minimally invasive fenestration), time (2 days, 1 month, 3 months, 1 year postoperatively), and time-treatment interaction, with results reported as least squares means and 95% confidence intervals. Robust standard errors and test statistics were calculated for the fixed effects. Appropriate comparisons were made within the mixed-effects model for repeated measures to compare least squares means between treatment groups at each time point and within each treatment group across time points. Considering the various etiologies of lumbar spinal stenosis such as disc degeneration, ligamentum flavum hypertrophy, and bone hyperplasia, this study will perform multivariate adjustments and subgroup analyses based on etiology. All analyses were conducted using R software version 4.3.3, primarily utilizing the lme4 and emmeans packages. A P-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with single-segment lumbar spinal stenosis through CT and MRI imaging combined with clinical symptoms;
* Symptoms in the lumbar region and lower extremities corresponding to the imaging findings;
* Patients who have not responded to three months of conservative treatment;
* Informed consent from family members regarding the surgical procedure and associated risks.

Exclusion Criteria:

* Patients with multi-segment lumbar disc herniation, malignant spinal tumors, spinal deformities, and other diseases.
* Patients with comorbidities such as cardiovascular diseases, cerebrovascular diseases, or those with mental abnormalities, communication difficulties, or other issues that may affect clinical evaluation.
* Patients with a history of previous lumbar surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index scores | 1 year postoperatively
  The maximum score is 100 points, and the minimum score is 0 points. The higher the score, the more severe the functional impairment.

SECONDARY OUTCOMES:
The Oswestry Disability Index scores | preoperatively, 1 day, 3 months, and 6 months postoperatively
  The maximum score is 100 points, and the minimum score is 0 points. The higher the score, the more severe the functional impairment.
Visual Analogue Score for lower limb pain/lumbar back pain | preoperatively, 1 day, 3 months, 6 months, and 1 year postoperatively
  The maximum score is 10 points, and the minimum score is 0 points. A higher score means a worse outcome and a more severe pain.
The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36 score) | preoperatively, 1 day, 3 months, 6 months, and 1 year postoperatively
  The scales was divided into 9 parts. For each part, the maximum score is 100 points, and the minimum score is 0 points. A higher score means the better outcome.
Dural sac cross-sectional area calculated from lumbar MRI | preoperatively and at 1 year postoperatively
  The Dural sac cross-sectional area (DCSA) refers to the two-dimensional area enclosed by the outer boundary of the dural sac as seen on imaging, typically measured in square millimeters (mm²). A reduced DCSA is often used to diagnose spinal stenosis.
  Anterior Boundary: The posterior longitudinal ligament and the vertebral body or intervertebral disc.
  Posterior Boundary: The inner surface of the ligamentum flavum or the posterior vertebral arch.
  Lateral Boundary: The inner walls of the pedicles or the edges of the vertebral foramen.
  These boundaries are identified on axial MRI imaging. The increase rate of the postoperative dural sac cross-sectional area at the last follow-up would be also calculated using Image J, which was defined as the [(postoperative dural sac cross-sectional area - preoperative dural sac cross-sectional area) / preoperative dural sac cross-sectional area].
Creatine kinase-MB (CK-MB) | preoperative and immediate postoperative
  preoperative and immediate postoperative changes in creatine kinase-MB (CK-MB)
Surgery time | Immediate postoperatively
Intraoperative blood loss | Immediate postoperatively
Surgical incision length | Immediate postoperatively
Postoperative hospital stay | Immediate postoperatively
Perioperative complication rate | Immediate postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Han S, Zeng X, Zhu K, Wu X, Shen Y, Han J, Lin A, Meng S, Zhang H, Li G, Liu X, Tao H, Ma X, Zhou C. Clinical Application of Large Channel Endoscopic Systems with Full Endoscopic Visualization Technique in Lumbar Central Spinal Stenosis: A Retrospective Cohort Study. Pain Ther. 2022 Dec;11(4):1309-1326. doi: 10.1007/s40122-022-00428-3. Epub 2022 Sep 3. PMID 36057015
- [Background] Katz JN, Zimmerman ZE, Mass H, Makhni MC. Diagnosis and Management of Lumbar Spinal Stenosis: A Review. JAMA. 2022 May 3;327(17):1688-1699. doi: 10.1001/jama.2022.5921. PMID 35503342
- [Background] Butcher NJ, Monsour A, Mew EJ, Chan AW, Moher D, Mayo-Wilson E, Terwee CB, Chee-A-Tow A, Baba A, Gavin F, Grimshaw JM, Kelly LE, Saeed L, Thabane L, Askie L, Smith M, Farid-Kapadia M, Williamson PR, Szatmari P, Tugwell P, Golub RM, Monga S, Vohra S, Marlin S, Ungar WJ, Offringa M. Guidelines for Reporting Outcomes in Trial Reports: The CONSORT-Outcomes 2022 Extension. JAMA. 2022 Dec 13;328(22):2252-2264. doi: 10.1001/jama.2022.21022. PMID 36511921
- [Background] Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, Coumans JV, Harrington JF, Amin-Hanjani S, Schwartz JS, Sonntag VK, Barker FG 2nd, Benzel EC. Laminectomy plus Fusion versus Laminectomy Alone for Lumbar Spondylolisthesis. N Engl J Med. 2016 Apr 14;374(15):1424-34. doi: 10.1056/NEJMoa1508788. PMID 27074067
- [Background] Forsth P, Olafsson G, Carlsson T, Frost A, Borgstrom F, Fritzell P, Ohagen P, Michaelsson K, Sanden B. A Randomized, Controlled Trial of Fusion Surgery for Lumbar Spinal Stenosis. N Engl J Med. 2016 Apr 14;374(15):1413-23. doi: 10.1056/NEJMoa1513721. PMID 27074066